CLINICAL TRIAL: NCT02072889
Title: Optimal Angle For Internal Jugular Cannulation
Brief Title: Optimal Neck Angle for Internal Jugular Cannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0220110074
Record Dates: First submitted 2014-02-10; First posted 2014-02-27 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Surgery
Keywords: Cardiac Surgery; Internal Jugular Cannulation; Optimal Neck Angle
MeSH Terms: interventions — Patient Positioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neck Angle Measures (Experimental): Subjects will position his/her neck in order to measure distance between the internal jugular and the carotid artery to determine if there is a maximal distance to target prior to cannulation
  Interventions: Other: Neck Angle

INTERVENTIONS:
Other: Neck Angle — Ultrasound guided measures of the neck of subjects undergoing cardiac surgery who need internal jugular vein cannulated
  Other Names: Position; Measurment; Distance

SUMMARY:
Measurements will be made between the internal jugular vein and the carotid artery using an ultrasound machine as the subjects is asked to move and position his or her neck in various positions.

It is hypothesized that by movements of the neck the investigators can maximize the distance between the internal jugular vein and the carotid artery to decrease inadvertent cannulation of the carotid artery to improve patient safety

DETAILED DESCRIPTION:
Patients will be asked to participate in this trial if they are scheduled for surgery and they will have their neck repositioned in several ways using an ultrasound machine to measure the distance between the internal jugular vein and the carotic artery to determine maximal distance in order to insert a catheter prior to surgery

ELIGIBILITY:
Inclusion Criteria:

Male and Females 18 years through 98 Scheduled for cardiac surgery Requires internal cannulation for their scheduled operative procedure -

Exclusion Criteria:

Individuals who refuse participation Subjects who already have had the internal jugular cannulated (line already present) History of carotid surgery History of Neck Surgery Individuals under 18 years of age

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Find Optimal Angle for internal jugular cannulation | Approximately 4 years
  Is there an angle to position ones neck which maximizes distances of carotid artery and internal jugular.

SECONDARY OUTCOMES:
Find Optimal Neck Angle | Approx 4 years
  Using the Ultrasound machine and having the subject position his neck measurements will be taken between the internal jugular and carotid artery to determine what angle may provide the maximal distance in order to safely cannulated the internal jugular

CONTACTS AND LOCATIONS:
Overall Officials: Vincent DeAngelis, MD, Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (1):
- Robert Wood Johnson University Hospital, New Brunswick, New Jersey, United States